CLINICAL TRIAL: NCT05495542
Title: Does "ShotBlocker" Affect Pain and Satisfaction During Diphtheria-Tetanus Vaccination in Pregnant Women? A Randomized Controlled Trial
Brief Title: The Effect of ShotBlocker on Injection Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bornova No. 25 Mevlana Family Health Center (Other)
Responsible Party: Principal Investigator, Merve Ince, Research Assistant, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 3023010044
Record Dates: First submitted 2022-08-05; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Pain; Intramuscular Injection
Keywords: diphtheria-tetanus vaccine; intramuscular injection; pain; pain management; patient satisfaction; pregnant woman
MeSH Terms: conditions — Pain; Agnosia; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The participants in the study and the researcher who evaluated the pain were blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shotblocker group (Experimental): In the ShotBlocker group, ShotBlocker was placed on the previously determined injection site before vaccination, and the vaccination was performed by holding it on the surface of the skin and pressing lightly with the fingertips. All vaccinations were carried out by an experienced nurse. ShotBlocker was removed after removing the needle.
  Interventions: Other: ShotBlocker
- Control group (No Intervention): In the control group, the steps of administering a normal intramuscular injection were used. Except for this, no additional method was used. All vaccinations were carried out by an experienced nurse.

INTERVENTIONS:
Other: ShotBlocker — ShotBlocker (Bionix, Toledo, OH) is one of the methods that can be used to reduce pain caused by IM injections. This small, flat, U-shaped plastic device used by holding it on the skin surface during injection did not have any side effects [5]. ShotBlocker has a surface of 2 mm thick with rounded nubs to stimulate the skin (Figure 1). The surface of the plastic device is placed on the skin just before the injection; there is a hole in the center where the injection is administered [6]. The rounded nubs on the surface of the plastic device do not damage the skin, these rounded nubs that create a slight pressure provide a warning for the Gate Control Theory [7]
  Arms: Shotblocker group

SUMMARY:
Shotblocker is an effective approach to reduce injection pain. Generally, injection pain has been studied in children, but reducing injection pain in adults is an important issue. This study investigates the effect of ShotBlocker on pain and satisfaction levels associated with diphtheria-tetanus vaccination in pregnant women.

The sample of this prospective, single-blind randomized controlled experimental study consists of 146 pregnant women registered to the Family Health Center between October 2018 and June 2019. Women were assigned to ShotBlocker and control groups with 73 women in each group. The women's pulse rate was taken one minute before the injection by the researcher. In the ShotBlocker group was used ShotBlocker. The control group used the steps of administering a normal intramuscular injection. The pain and satisfaction related to the injection were evaluated using the Visual Analog Scale and Visual Patient Satisfaction Scale after the vaccination. Pulse rates of the women were taken again by the researcher one minute after the injection.

DETAILED DESCRIPTION:
As the rate of vaccination increases, preventable diseases and their negative effects decrease; Nevertheless, the significance of vaccine-related side effects is increasing. The most prevalent complications in vaccine applications are local reactions such as pain, swelling, and erythema at the injection site. The most frequent pain in these reactions develops after diphtheria-tetanus vaccine in which aluminum is used as an adjuvant. Diphtheria-tetanus vaccine is generally administered to the deltoid region by intramuscular injection (IM), and most pregnant women complain about the pain that they experience during and after administration of diphtheria-tetanus vaccine. Nurses have a great responsibility in reducing and eliminating the pain felt by patients during operations. The success of pain management is related to nurses' knowledge and skills. If the pain that an individual will feel due to the piercing of the skin with a needle during intramuscular injection application is decreased or reduced to minimum, the anxiety and fear that the person will experience may abate. Therefore, to reduce pain and anxiety in individuals during injection; nurses use many non-pharmacological methods. ShotBlocker (Bionix, Toledo, OH) is one of the methods that can be used to reduce pain caused by IM injections. This small, flat, U-shaped plastic device used by holding it on the skin surface during injection did not have any side effects. ShotBlocker has a surface of 2 mm thick with rounded nubs to stimulate the skin. The surface of the plastic device is placed on the skin just before the injection; there is a hole in the center where the injection is administered. The rounded nubs on the surface of the plastic device do not damage the skin, these rounded nubs that create a slight pressure provide a warning for the Gate Control Theory. ShotBlocker's mechanism of action is thought to reduce pain by stimulating nerve endings faster with pressure of rounded nubs on the device. This stimulation decreases pain by blocking pain signals temporarily during injections and by inhibiting the central nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and understand Turkish
* Those who volunteered to participate in the study and received written consent
* 18 years old and over
* Those with tetanus+diphtheria vaccination prescription/demand
* No vision-hearing-speech problems
* No secondary cause of acute pain other than intramuscular injection.
* Pregnant women who do not have a physical disability (burn, absence or amputation of an extremity, contracture, tissue necrosis, etc.) for injection into the deltoid muscle.

Exclusion Criteria:

* Pregnant women who cannot speak Turkish
* Younger than 18
* Pregnant women who do not want to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women were included in the study.
Enrollment: 146 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | 6 month
  The VAS is used to assess the severity of acute pain. It is mostly a horizontal or vertical line 100 mm long, starting with "no pain" and ending with "unbearable pain". It is used to convert some values that cannot be measured numerically to a numerically usable form [10].

SECONDARY OUTCOMES:
Visual patient satisfaction scale | 6 month
  The visual patient satisfaction scale combines the characteristics of the well-known VAS. At one end of the scale is the phrase "I am not satisfied at all", and at the other end is the phrase "I am very satisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Leyla KHORSHID, Professor, Principal Investigator — khorshidleyla@gmail.com
Locations (1):
- Merve, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Drago LA, Singh SB, Douglass-Bright A, Yiadom MY, Baumann BM. Efficacy of ShotBlocker in reducing pediatric pain associated with intramuscular injections. Am J Emerg Med. 2009 Jun;27(5):536-43. doi: 10.1016/j.ajem.2008.04.011. PMID 19497458
- [Result] Romano CL, Cecca E. A new method to reduce pin-prick pain of intra-muscular and subcutaneous injections. Minerva Anestesiol. 2005 Oct;71(10):609-15. English, Italian. PMID 16163151
- [Result] Cobb JE, Cohen LL. A randomized controlled trial of the ShotBlocker for children's immunization distress. Clin J Pain. 2009 Nov-Dec;25(9):790-6. doi: 10.1097/AJP.0b013e3181af1324. PMID 19851160